CLINICAL TRIAL: NCT01509365
Title: Evaluation the Effect of the Double Maintenance Dose of Clopidogrel Versus Single Dose in Patients With Coronary Artery Disease With a BMI ≥ 27 kg.m-2
Brief Title: Effect of Platelet Inhibition According to Clopidogrel Dose in Patients With Body Mass Index ≥ 27
Acronym: PLATO-dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Collaborators: University Hospital Fattouma Bourguiba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03 PID 11
Record Dates: First submitted 2012-01-09; First posted 2012-01-13 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2014-10

CONDITIONS: Cardiovascular Disease; Overweight
Keywords: cardiovascular disease; maintenance dose; clopidogrel; overweight; antiplatelet agents
MeSH Terms: conditions — Cardiovascular Diseases; Overweight | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sensible (No Intervention): Patients who show adequate response to loading dose of clopidogrel and receive standard 1x75 mg clopidogrel for at least 7 days.
- simple dose (Active Comparator): Patients who show suboptimal response to loading dose of clopidogrel and receive 1x75 mg clopidogrel for 1 month followed by standard 75 mg clopidogrel for 3 months to one year.
  Interventions: Drug: clopidogrel
- double dose (Experimental): Patients who show suboptimal response to loading dose of clopidogrel and receive 1x150 mg clopidogrel for 1 month followed by standard 75 mg clopidogrel for 3 months to one year.
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: clopidogrel — 2 tablets of 75 mg clopidogrel for one month followed by standard 75 mg clopidogrel for 3 months to one year.
  Arms: double dose
Drug: clopidogrel — 1 tablet of 75 mg clopidogrel for one month followed by standard 75 mg clopidogrel for 3 months to one year.
  Arms: simple dose

SUMMARY:
The purpose of the study is to determine whether administration of 150 mg clopidogrel is effective in reducing the one-year incidence of thromboischemic events in patients with high on-clopidogrel platelet reactivity compared to 75 mg clopidogrel in the patient population overweight or obese with a body mass index (BMI) ≥ 27 kg.m-2.

DETAILED DESCRIPTION:
The goal is to evaluate the effect of the double maintenance dose of clopidogrel versus single dose in patients with proven coronary and with BMI ≥ 27 kg.m-2 1 - Biologically: study and compare the respective effects of the double dose and single dose of clopidogrel on platelet aggregation.

2 - Clinically: to study and compare the cardiovascular events and adverse effects depending on the dose of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* Old (e) of more than 20 years
* BMI ≥ 27kg.m-2
* Patients hospitalized for acute coronary syndrome (Whatever the ST segment and troponin dosage)
* Patients with proven coronary candidates for treatment with Clopidogrel (who received a loading dose of 600mg over 2 hours or treated with 75 mg/day or 150mg / day of clopidogrel for longer than 7 days)

Exclusion Criteria:

* Patients unwilling.
* Patient participating in another study.
* Patients with cardiogenic shock
* Patient on anti GpIIbIIIa or stopped less than 72 hours before the test aggregability
* Patients scheduled for surgery in less than 6 months
* ischemic stroke older than 6 weeks.
* History of hemorrhagic stroke (any time)
* Patients on or candidates for AVK
* Patients with a different anti ADP (ticlopidine, prasugrel)
* Patients with an indication against clopidogrel (side effects, bleeding ...)
* Thrombocytopenia < 100000/mm3
* anemia (Ht < 30%)
* Thrombocythaemia (Ht > 52%)
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Cardiac death or non-fatal myocardial infarction or ischemia-driven target vessel revascularisation | 6 months

SECONDARY OUTCOMES:
ADP-induced platelet aggregation assessed by VerifyNow test | 7 days after selection of patients

CONTACTS AND LOCATIONS:
Overall Officials: Faouzi Maatouk, MD, Study Chair — hospital Fattouma Bourguiba; Khaldoun Ben Hamda, MD, Principal Investigator — Hospital Fattouma Bourguiba; Sonia Hamdi, MD, Principal Investigator — Hospital Fattouma Bourguiba; Mohsen Hassine, Principal Investigator — Hospital Fattouma Bourguiba
Locations (1):
- cardiology department, hospital Fattouma Bourguiba, Monastir, Monastir Governorate, Tunisia